CLINICAL TRIAL: NCT00737425
Title: Evaluation of Safety and Efficacy of the PainShield Device for the Treatment of Subjects Who Underwent Laparoscopic-Assisted Abdominal Surgery
Brief Title: Safety and Efficacy Study of Pain Shield Device to Treat Subjects Following Laparoscopic-Assisted Abdominal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Nanovibronix (Industry)
Responsible Party: Prof Petachia Reissman, Head of Surgery Department, Shaare Zedek Medical Center, Jerusalem, Israel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NV-PS-02-001
Record Dates: First submitted 2008-08-17; First posted 2008-08-19 (Estimated); Last update posted 2008-10-28 (Estimated); Status verified 2008-10

CONDITIONS: Wounds
Keywords: laparoscopic-assisted surgery; abdominal; pain relief; wound healing; low intensity ultrasound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Active Comparator)
  Interventions: Device: PainShield
- 2 (Sham Comparator)
  Interventions: Device: Sham PainShield

INTERVENTIONS:
Device: PainShield
  Arms: 1
Device: Sham PainShield
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of PainShield device, based on ultrasound technology, for postoperative pain relief and wound healing following a laparoscopic-assisted abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject's Age ≥ 18
* Subject is able, agrees and signs the Informed Consent Form
* Subject requires laparoscopic-assisted abdominal surgery
* Incision size following the laparoscopy between 4-7 cm

Exclusion Criteria:

* Epidural analgesia
* IV PCA
* Subject has any condition, which precludes compliance with study and/or device instructions
* Subject is currently participating in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-09

PRIMARY OUTCOMES:
Pain and discomfort will be measured using appropriate validated questionnaires. | Pain assessment will be performed daily

SECONDARY OUTCOMES:
Infections will be assessed by concomitant antibiotic intake | Concomitant medications will be assessed daily

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel